CLINICAL TRIAL: NCT07113821
Title: Biceps Tenodesis Alone Versus Biceps Tenodesis and Labrum Repair in Superior Labrum Anteroposterior ( SLAP) From Type II to Type IV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous Fouad Mohamed, Resident of orthopaedic and trauma surgery Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLAP lesion from type II to IV
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: SLAP Lesion

STUDY DESIGN:
Intervention Model Description: 2 parallel groups selected by Randomisation
Who Masked: Outcomes Assessor
Masking Description: Aim of this study is comparing outcome results of biceps tenodesis alone versus biceps tenodesis and labrum repair in superior labrum anteroposterior ( SLAP) from type II to type IV
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biceps tenodesis alone (Other)
  Interventions: Procedure: Biceps tenodesis alone
- Biceps tenodesis and labrum repair (Other)
  Interventions: Procedure: Biceps tenodesis and labrum repair

INTERVENTIONS:
Procedure: Biceps tenodesis alone — Biceps tenodesis in superior labrum anteroposterior lesion from type II to type IV
  Arms: Biceps tenodesis alone
Procedure: Biceps tenodesis and labrum repair — Biceps tenodesis and labrum repair by anchors in superior labrum anteroposterior lesion from type II to type IV
  Arms: Biceps tenodesis and labrum repair

SUMMARY:
Biceps Tenodesis Alone Versus Biceps Tenodesis and Labrum Repair in Superior Labrum Anteroposterior ( SLAP) From Type II to Type IV

DETAILED DESCRIPTION:
A SLAP (Superior Labrum Anterior to Posterior) lesion is a specific type of shoulder injury that involves damage to the superior labrum, which is the cartilage rim around the socket of the shoulder joint. This type of injury typically occurs at the long head of the biceps tendon attaches to the labrum. The patient may feel pain, popping sensations and decreased range of motion in the shoulder.1 SLAP lesions are occurring in younger individuals,who playing sports that require repetitive overhead motions and presenting in individuals who have shoulder trauma injury,such as a fall or a direct blow to the shoulder.5There are four main types of SLAP lesions: in this research including from type II to type IV . SLAP type II is characterized by superior part of the labrum , along with the biceps tendon is detached from the glenoid . SLAP type III is characterized by bucket handle tear of the superior labrum , where a piece of the labrum detaches and flips into the shoulder . SLAP type IV is characterized by a bucket-handle tear of the superior labrum that extends into the biceps tendon. The prevalence of SLAP lesions as a cause of shoulder pain is estimated to be around 6-26% in the general population. 2,3,4,5,6Treatment of SLAP lesion is biceps tenodesis which was recently described, used suture anchor for fixation the biceps tendon to proximal humerus to obtain the stability of glenohumeral muscle. Fixation methods include tenodesis through a bone tunnel which have a role in pain relief and maintain biceps muscle strength and have a role in preventing cramping.7,8 Recently treatment of SLAP lesion is repairing the labrum using suture anchors with Biceps tenodesis.1 This study prepared to compare the results of biceps tenodesis alone Versus biceps tenodesis and labrum repair in superior labrum anteroposterior (SLAP) Lesion from type II to type IV .

ELIGIBILITY:
Inclusion Criteria:

* Traumatic and degenerative etiology.
* No shoulder deformity .
* No inflammatory joint disorders.
* Type of the SLAP is SLAP lesion from type II to type IV

Exclusion Criteria:

* History of the disease.
* Bilateral shoulder.
* DM .
* Epilepsy .
* psychological disturbance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome by American shoulder elbow score | 12 months
  Examination of the patients and ask them about their pain degree and record the results
VAS score | 12months
  Examination of the patients and ask them about their pain degree and record the results

REFERENCES:
- See also: American Academy of Orthopaedic Surgeons. (2018). SLAP Tears. Retrieved from https://orthoinfo.aaos.org/en/diseases--conditions/slap-tears/. — http://orthoinfo.aaos.org/en/diseases--conditions/slap-tears/